CLINICAL TRIAL: NCT01451398
Title: A Phase 3, Multicenter, Double-blind, Placebo-controlled, Randomized, Clinical Trial Evaluating the Efficacy and Safety of Prandial Technosphere® Insulin Inhalation Powder Versus Technosphere Inhalation Powder in Insulin Naïve Subjects With Type 2 Diabetes Mellitus Poorly Controlled With Oral Antidiabetic Agents Over a 24 Week Treatment Period
Brief Title: Comparison of Technosphere® Insulin Versus Technosphere Powder (Placebo) in Insulin-Naive Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKC-TI-175; Affinity2
Record Dates: First submitted 2011-10-07; First posted 2011-10-13 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TI inhalation powder (Experimental): Technosphere® Insulin powder administered via the Gen2 inhaler added to 2 or more stable OADs
  Interventions: Drug: Technosphere® Insulin
- Technosphere powder (Placebo Comparator): Technosphere powder (with no insulin) administered via the Gen2 inhaler added to 2 or more stable OADs
  Interventions: Drug: Technosphere Powder

INTERVENTIONS:
Drug: Technosphere® Insulin — Technosphere® Insulin Inhalation Powder
  Arms: TI inhalation powder
Drug: Technosphere Powder — Placebo Comparator
  Arms: Technosphere powder

SUMMARY:
Insulin-naive subjects with Type 2 Diabetes Mellitus who are sub-optimally controlled on either maximum tolerated dose of metformin or maximum tolerated dose of metformin plus one or two other oral anti-diabetic medications will have either Prandial Technosphere® Insulin or Technosphere Powder (placebo) added to their oral antidiabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > or = to 7.5% and < or = to 10.0%
* Body mass index (BMI) < or = to 45 kg/m2
* Non smoker for at least 6 months before Screening
* Clinical diagnosis of type 2 diabetes mellitus for more than 12 months
* Currently receiving as diabetes treatment only metformin or 2 or more OADs and on stable doses for at least 3 months before enrollment

  * Subjects receiving metformin must be on at least 1.5gm daily, or up to the maximum tolerated dose
  * Subjects treated with a sulfonylurea must be on at least 50% of the total maximum approved dose for a given agent
  * Subjects receiving a DPP-4 inhibitor must receive the maximum approved dose specific for that agent
  * Metiglinide and alpha-glucoside inhibitors must be taken at the highest tolerated dose within the approved dose range
* No previous or current treatment with insulin, except during an acute illness, gestational diabetes, or at time of initial diagnosis of diabetes
* Forced expiratory volume in one second (FEV1) > or = to 70% Third National Health and Nutrition Examination Survey (NHANES III) predicted
* Forced vital capacity (FVC) > or = to 70% NHANES III predicted
* Forced expiratory volume in one second as a percentage of forced vital capacity (FEV1/FVC) > or = to NHANES III lower limit of normal (LLN)

Exclusion Criteria:

* History of chronic obstructive pulmonary disease (COPD), clinically proven asthma, or any other clinically important pulmonary disease (eg, pulmonary fibrosis)
* Any clinically significant radiological findings on screening chest x-ray
* Use of medications for asthma, COPD, or any other chronic respiratory conditions
* Evidence of serious complications of diabetes (proliferative retinopathy, autonomic neuropathy with symptoms of gastroparesis or cardiac arrhythmia; sensory neuropathy that makes manipulation of the Gen2C inhaler difficult)
* Renal disease or renal dysfunction
* Significant cardiovascular dysfunction or history thereof within 12 months of screening; serious arrhythmia, treatment with medications to control/treat arrhythmias; myocardial infarction; cardiac surgery; history of valvular heart disease
* Previous or current use of amiodarone
* Treatment with glucagon-like peptide-1 (GLP-1) analogs, thiazolidinediones (TZD), or weight loss drugs (eg, sibutramine, orlistat) within 3 months of screening
* History of pulmonary embolism or deep venous thrombosis in the 12 months before Screening
* History of recent blood transfusion (within previous 3 months) or diagnosis of hemoglobinopathies that may affect HbA1c measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (44):
  - Anaheim, California
  - Huntington Beach, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Tustin, California
  - West Hills, California
  - Hialeah, Florida
  - Hollywood, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - North Miami Beach, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Dunwoody, Georgia
  - Lawrenceville, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Baton Rouge, Louisiana
  - Edina, Minnesota
  - City of Saint Peters, Missouri
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Clifton, New Jersey
  - Hackensack, New Jersey
  - Paramus, New Jersey
  - Flushing, New York
  - New Hyde, New York
  - Greenville, North Carolina
  - Perrysburg, Ohio
  - Portland, Oregon
  - Greer, South Carolina
  - Memphis, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Magna, Utah
  - Renton, Washington
  - Wenatchee, Washington
- Brazil (2):
  - Porto Alegre
  - São Paulo
- Russia (7):
  - Kemerovo
  - Leningrad Region
  - Moscow
  - Petrozavodsk
  - Saint Petersburg
  - Smolensk
  - Yaroslavl
- Ukraine (6):
  - Kharkiv, UKR
  - Kiev, UKR
  - Kyiv, UKR
  - Odesa, UKR
  - Vinnytsia, UKR
  - Kiev

REFERENCES:
- [Derived] Rosenstock J, Franco D, Korpachev V, Shumel B, Ma Y, Baughman R, Amin N, McGill JB; Affinity 2 Study Group. Inhaled Technosphere Insulin Versus Inhaled Technosphere Placebo in Insulin-Naive Subjects With Type 2 Diabetes Inadequately Controlled on Oral Antidiabetes Agents. Diabetes Care. 2015 Dec;38(12):2274-81. doi: 10.2337/dc15-0629. Epub 2015 Aug 7. PMID 26253730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient enrolled November 2011. Multi-national trial conducted in US, Russia, Ukraine and Brazil
Pre-assignment Details: 6 week Screening Period prior to OAD run-in period. 1379 Screened /539 Eligible of which 535 entered the run-in period. 439 met randomization criteria at end of run-in of which 353 were randomized.
Groups:
- TI Inhalation Powder + OADs: Technosphere Insulin powder administered via the Gen2 inhaler added to 2 or more stable Oral Antidiabetic Drugs (OADs), doses individualized for each patient
- Technosphere Powder: Technosphere powder (with no insulin) administered via the Gen2 inhaler added to 2 or more stable Oral Antidiabetic Drugs (OADs), doses individualized for each patient
Period: Overall Study
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Started | 177 | 176
Completed | 150 | 139
Not Completed | 27 | 37
Not completed — Adverse Event | 7 | 9
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 10 | 14
Not completed — Lost to Follow-up | 6 | 4
Not completed — Non-compliance with study drug | 1 | 3
Not completed — Non-compliance with protocol | 1 | 1
Not completed — Moved out of country | 0 | 1
Not completed — Adverse Event + Elevated Fasting Glucose | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder | Total
Number analyzed (Participants) | 177 | 176 | 353
Age, Customized [Number; unit: participants]
  18-30 years | 1 | 0 | 1
  31-49 years | 37 | 33 | 70
  50-64 years | 102 | 110 | 212
  >=65 years | 37 | 33 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 102 | 197
  Male | 82 | 74 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 17 | 38
  White | 151 | 155 | 306
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 41 | 84
  Not Hispanic or Latino | 134 | 135 | 269
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 88 | 87 | 175
  Brazil | 15 | 14 | 29
  Ukraine | 19 | 19 | 38
  Russian Federation | 55 | 56 | 111
Duration of Diabetes [Mean (Full Range); unit: years] | 9.7 [1.1 to 34.7] | 9.2 [1.0 to 28.8] | 9.5 [1.0 to 34.7]
Weight [Mean (Full Range); unit: kg] | 90.2 [54.0 to 142.3] | 90.8 [58.0 to 136.6] | 90.5 [54.0 to 142.3]
BMI [Mean (Full Range); unit: kg/m^2] | 31.8 [21.6 to 44.6] | 32.4 [21.1 to 44.4] | 32.1 [21.1 to 44.6]
Fasting Plasma Glucose (FPG) [Mean (Full Range); unit: mg/dL] | 179.1 [49 to 306] | 177.2 [54 to 316] | 178.2 [49 to 316]
HbA1c [Mean (Full Range); unit: Percent of hemoglobin] | 8.26 [6.6 to 10.1] | 8.35 [5.1 to 10.9] | 8.31 [5.1 to 10.9]
Oral Anti-Diabetic Drug (OAD) Type [Number; unit: participants]
  Metformin Only | 42 | 40 | 82
  Metformin + Sulfonylurea | 114 | 115 | 229
  Metformin + DPP-4 Inhibitor | 9 | 9 | 18
  Metformin + 1 or more OADs not specified above | 9 | 9 | 18
  2 or more OADs (not including Metformin) | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in HbA1c
Description: Efficacy as measured by change in glycated hemoglobin (HbA1c) at Week 24
Time Frame: Baseline to Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
percentage of hemoglobin | -0.82 (0.061) | -0.42 (0.062)
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Change in HbA1c = Baseline HbA1c + Region + Pooled OAD Strata + Visit + Treatment + (Treatment*Visit), using AR(1) variance/covariance structure; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.57 to -0.23]

2. Secondary Outcome: Proportion of Responders Achieving HbA1c <= 7.0%
Description: Efficacy as measured in proportion of subjects achieving HbA1c < or = to 7.0%
Time Frame: Week 24
Population: Full analysis set for subjects with available data at Week 24
Measure: Number; unit: percentage of participants
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 151 | 142
percentage of participants | 37.7 | 19.0
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Model: Treatment + Pooled OAD Stratum + Region + Baseline HbA1c; Odds Ratio (OR) = 2.726, 95% CI 2-sided [1.55 to 4.80]

3. Secondary Outcome: Proportion of Responders Achieving HbA1c <= 6.5%
Description: Efficacy as measured in proportion of subjects achieving HbA1c < or = to 6.5% at Week 24
Time Frame: Week 24
Population: Full analysis set for subjects with available data at Week 24
Measure: Number; unit: percentage of participants
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 151 | 142
percentage of participants | 15.9 | 4.2
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p = 0.0021, Regression, Logistic; Model: Treatment + Pooled OAD Stratum + Region + Baseline HbA1c; Odds Ratio (OR) = 4.361, 95% CI 2-sided [1.70 to 11.17]

4. Secondary Outcome: FPG Change From Baseline to Week 24
Description: Efficacy as measured by mean change in fasting plasma glucose (FPG)
Time Frame: Baseline to Week 24
Population: Full analysis set for subjects with data at both Baseline and at Week 24
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 139 | 128
mg/dL | -11.20 (3.776) | -3.78 (3.864)
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p = 0.1698, Mixed Models Analysis; Model: FPG = Baseline FPG + Region + Pooled OAD Stratum + Visit + Treatment + (Treatment * Visit) Variance/Covariance Matrix is Autoregression 1; Mean Difference (Net) = -7.42, 95% CI 2-sided [-18.03 to 3.18], Standard Error of Mean 5.400

5. Secondary Outcome: Proportion of Subjects Requiring Rescue Therapy
Time Frame: Baseline to Week 24
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
percentage of participants | 6.8 | 9.7

6. Secondary Outcome: Time to Rescue
Description: Time from Week 0 (baseline) to initiation of rescue therapy (up to a maximum of 24 weeks/end of treatment) for subjects not responding to treatment
Time Frame: Baseline to Week 24
Population: Full analysis set
Measure: Median (Full Range); unit: Days
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
Days | 95 [22 to 141] | 85 [28 to 160]

7. Secondary Outcome: FEV1 Change From Baseline to Week 24
Description: Forced Expiratory Volume in 1 second - change from baseline to week 24
Time Frame: Baseline to Week 24
Population: Full analysis set for patients with data at both Baseline and at Week 24
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 141 | 122
Liters | -0.13 (0.175) | -0.04 (0.147)
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; Mixed Models Analysis; FEV1 = Baseline FEV1 + Age + Gender + Race + Height + Visit + Treatment + (Treatment*Visit); Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.12 to -0.05], Standard Deviation 0.018

8. Secondary Outcome: Incidence of Total Hypoglycemia
Description: Hypoglycemia, defined as blood glucose <= 70 mg/dL or in absence of blood glucose, symptoms that are resolved by the administration of carbohydrates.
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
percentage of participants | 67.8 | 30.7

9. Secondary Outcome: Incidence of Severe Hypoglycemia
Description: Severe Hypoglycemia defined as: Requiring 3rd party assistance.
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
percentage of participants | 5.1 | 1.7

10. Secondary Outcome: Total Hypoglycemia Event Rate
Description: Number of Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: Events/Subject-Month
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
Events/Subject-Month | 1.16 | 0.50
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p < 0.0001, Negative binomial regression; Model: Treatment + Region + OAD Stratum + Exposure Time

11. Secondary Outcome: Severe Hypoglycemia Event Rate
Description: Number of Severe Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Number; unit: Events/100 Subject-Month
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
Events/100 Subject-Month | 2.37 | 0.60
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p = 0.2024, Negative Binomial Regression; Model: Treatment + Region + OAD Stratum + Exposure Time

12. Secondary Outcome: Mean 7-point Glucose Baseline Values
Description: Mean 7-point self-monitored glucose at baseline
Time Frame: Baseline
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 177 | 176
mg/dL
  Before Breakfast | 178.5 (37.58) | 182.2 (40.50)
  After Breakfast | 212.8 (51.01) | 219.9 (51.77)
  Before Lunch | 176.7 (49.58) | 183.6 (53.76)
  After Lunch | 197.0 (46.94) | 209.1 (44.37)
  Before Dinner | 176.8 (41.81) | 187.6 (50.04)
  After Dinner | 205.2 (48.72) | 211.2 (50.44)
  Bedtime | 203.3 (50.55) | 203.8 (46.52)

13. Secondary Outcome: Mean 7-point Glucose Week 24 Values
Description: Mean 7-point self-monitored blood glucose at Week 24
Time Frame: Week 24
Population: Full analysis set for patients with data at Week 24
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 150 | 139
mg/dL
  Before Breakfast | 156.6 (30.80) | 160.9 (36.7)
  After Breakfast | 170.3 (44.23) | 194.7 (50.02)
  Before Lunch | 152.4 (48.13) | 163.4 (49.8)
  After Lunch | 158.0 (42.79) | 183.8 (47.73)
  Before Dinner | 157.4 (49.34) | 164.7 (40.60)
  After Dinner | 164.3 (44.84) | 188.5 (43.93)
  Bedtime | 163.0 (42.66) | 178.7 (44.50)

14. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight from Baseline to Week 24
Time Frame: Baseline to Week 24
Population: Full analysis set for patients with data at both Baseline and at Week 24
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | TI Inhalation Powder + OADs | Technosphere Powder
Number analyzed (Participants) | 152 | 142
kg | 0.49 (0.333) | -1.13 (0.347)
Statistical Analysis 1: Comparison: TI Inhalation Powder + OADs vs Technosphere Powder; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [0.90 to 2.34], Standard Error of Mean 0.365 — Model: Baseline Weight + Change in HbA1c at Week 24 + Region + OAD Stratum + Treatment

ADVERSE EVENTS:
Time Frame: 24 Weeks
Groups:
- TI Inhalation Powder: Technosphere® Insulin powder administered via the Gen2 inhaler added to 1 - 3 stable OADs
  Technosphere® Insulin: Technosphere® Insulin Inhalation Powder
- Technosphere Powder: technosphere powder (with no insulin) administered via the Gen2 inhaler added to 1 - 3 stable OADs
  Technosphere Powder: Placebo Comparator
Arm/Group | TI Inhalation Powder | Technosphere Powder
Serious Adverse Events (participants affected / at risk) | 5/177 | 9/176
Other Adverse Events (participants affected / at risk) | 108/177 | 82/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI Inhalation Powder (N=177) | Technosphere Powder (N=176)
Angina Pectoris (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 0
Skull Malformation (Congenital, familial and genetic disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Heart Rate Decreased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischemic Stroke (Nervous system disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI Inhalation Powder (N=177) | Technosphere Powder (N=176)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 35
Nasopharyngitis (Infections and infestations) | 15 | 8
Influenza (Infections and infestations) | 10 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Headache (Nervous system disorders) | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Urinary Tract Infection (Infections and infestations) | 6 | 2
Bronchitis (Infections and infestations) | 5 | 7
Nausea (Gastrointestinal disorders) | 4 | 0
Oedema Peripheral (General disorders) | 4 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 2 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.